CLINICAL TRIAL: NCT00835380
Title: A Phase III Open-Label Study of Immunogenicity, Safety, and Tolerability of 2 Doses of VAQTA™ (Formalin, Inactivated, Alum-Adjuvanted Hepatitis A Vaccine) in Healthy Children 12 to 23 Months of Age
Brief Title: A Study of 2 Doses of VAQTA™ in Healthy Children 12 to 23 Months of Age (V251-069)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V251-069; 2009_531
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2010-01-11 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Hepatitis A Virus Infection
MeSH Terms: interventions — Hepatitis A Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): VAQTA™
  Interventions: Biological: Hepatitis A Vaccine, Purified Inactivated (VAQTA™)

INTERVENTIONS:
Biological: Hepatitis A Vaccine, Purified Inactivated (VAQTA™) — Subjects will be given a 25-U/0.5 mL intramuscular injections of VAQTA™ at Day 1 and Month 6.
  Other Names: VAQTA™

SUMMARY:
This study will demonstrate the immunogenicity and evaluate the safety/tolerability of the vaccine in Chinese children between 12 and 23 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese children 12 to 17 months old at receipt of the first study vaccination

Exclusion Criteria:

* Subject is Hepatitis A virus antibody positive at screening or has a history of Hepatitis A infection
* Subject has a fever 72 hours prior to first injection
* Subject has already been vaccinated for Hepatitis A
* Subject is allergic to aluminum, formaldehyde, sodium borate, latex, or any component of the vaccine
* Subject has received inactivated vaccines within 14 days of screening or live vaccines within 30 days of screening

Ages: 12 Months to 23 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 114 subjects were enrolled for vaccination screening. Subject eligibility was reviewed according to the inclusion/exclusion criteria, and blood samples were collected for HAV (hepatitis A virus) antibody and ALT (alanine aminotransferase) testing. Finally 80 HAV-susceptible subjects with normal ALT were administered vaccines at the Day 1
Groups:
- VAQTA™: Subjects be given a 25-U/0.5-ml intramuscular injection of VAQTA™ at the Day 1 and Month 6 visits respectively.
Period: Overall Study
Arm/Group | VAQTA™
Started | 80
Completed | 78
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | VAQTA™
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Months] | 14.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 43
Body Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 35.56 (0.31)
Pulse [Mean (Standard Deviation); unit: Beats per minute (BPM)] | 80.05 (5.04)

OUTCOME MEASURES:

1. Primary Outcome: Hepatitis A Virus (HAV) Seroconversion Rate, i.e. the Percentage of Subjects Who Were Seronegative at Baseline and Developed Seropositive at Month 7 After Administration of a 2-dose Regime of Vaccines.
Description: Seroconversion rate = (number of subjects with seronegative at baseline and developed seropositive at Month 7)/(number of subjects with seronegative at baseline regardless HAV serum status at Month 7). Measure serum HAV (hepatitis A virus) antibody at Day 0 prior to vaccination and at Month 7 after administration of a 2-dose regimen of vaccines.
  HAV antibody titers were determined by Wantai ELISA kit for serum antibody response to HAV. Seropositive was defined as HAV antibody titer ≥ 50 mIU/mL. Seronegative was defined as HAV antibody titer < 50 mIU/mL.
Time Frame: Collect blood sample for HAV antibody testing at Day 0 prior to vaccination, and Month 7 (4 weeks after administration of a 2-dose regimen of vaccines at Month 6)
Population: Per-protocol population, defined as all HAV-susceptible subjects who completed the vaccination regimen within acceptable day ranges, had 2 valid serology results on Day 0 and Month 7, and met all inclusion/exclusion criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | VAQTA™
Number analyzed (Participants) | 70
Percentage of Participants
  Seronegative at Month 7 | 2
  Seropositive at Month 7 | 68
Statistical Analysis 1: Comparison: VAQTA™; Test type: Superiority or Other; Seroconversion Rate = 99, 95% CI [89 to 99]

2. Secondary Outcome: Serious Adverse Experiences and Systemic Adverse Experiences Occurring Within 14 Days After Each Vaccination, and Injection-site Complaints Occurring Day 1 Through Day 5 After Each Vaccination
Description: All adverse experiences were collected from the time the consent form was signed through 14 days following the first vaccination(s) and from the time of the second vaccination through 14 days thereafter. The parent/legal guardian of each participant were requested to record injection-site adverse experiences and monitor the subject's temperature daily on the Vaccination Report Card for Day 1 thereafter for 4 additional calendar days, and record all systemic adverse experiences that occur during the 14-day period after each injection.
Time Frame: For serious adverse experiences and systemic adverse experiences: 14 days follow-up after each dose of vaccination; For injection-site adverse experiences: 5 days follow-up after each dose of vaccination
Population: Safety population, defined as all subjects who were vaccinated at least one dose and had safety follow-up data
Measure: Number; unit: participants
Arm/Group | VAQTA™
Number analyzed (Participants) | 80
participants
  Serious adverse experiences | 0
  Injection-site adverse experiences | 10
  Systemic adverse experiences | 54

ADVERSE EVENTS:
Arm/Group | VAQTA™
Serious Adverse Events (participants affected / at risk) | 0/80
Other Adverse Events (participants affected / at risk) | 56/80
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VAQTA™ (N=80)
Injection site redness (General disorders) | 5 (6)
Injection site pain (General disorders) | 5 (6)
Injection site induration (General disorders) | 4 (4)
Injection site swelling (General disorders) | 4 (4)
Injection site pruritus (General disorders) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1)
Fidgety (Nervous system disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 15 (16)
Vomiting (Gastrointestinal disorders) | 3 (3)
Inappetency (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 1 (1)
Coughing (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 16 (28)
Bronchopenumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic reaction (General disorders) | 2 (2)
Fever (General disorders) | 34 (38)
Fatigue (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.